CLINICAL TRIAL: NCT05792462
Title: Efficacy and Safety of Baricitinib in Neuromyelitis Optica Spectrum Disorders
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University General Hospital (Other)
Collaborators: Tang-Du Hospital (Other); The Second Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Qiang Liu, Professor of Department of Neurology, Tianjin Medical University General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB2023-YX-012-01
Record Dates: First submitted 2023-03-18; First posted 2023-03-31 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: NMO Spectrum Disorder
MeSH Terms: conditions — Neuromyelitis Optica | interventions — baricitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Baricitinib (Experimental): Baricitinib will be taken orally with a dose of 2mg once daily until the disease relapses or week 48, with a final evaluation at week 52.
  Interventions: Drug: Baricitinib

INTERVENTIONS:
Drug: Baricitinib — Baricitinib will be taken orally with a dose of 4mg once daily until the disease relapses or week 48, with a final evaluation at week 52.

SUMMARY:
Neuromyelitis Optica Spectrum Disorders (NMOSD) is associated with a pathological humoral immune response against the aquaporin-4(AQP-4) water channel. Baricitinib is an oral Janus kinase (JAK)1/JAK2 inhibitor that blocks the upregulated JAK-STAT pathway in patients with neuroimmune disorders, which is important in bone marrow regulation of B cell proliferation and differentiation. Baricitinib may benefit some patients with NMOSD due to the important role of B cells in the pathogenesis of NMOSD. Clinical trials may be needed to observe its efficacy and safety.

DETAILED DESCRIPTION:
The investigators primarily aim to observe the number of attacks from initiation of baricitinib treatment.

The secondary outcomes are to determine: The safety profile of baricitinib in participants with NMO and whether baricitinib improves Expanded Disability Status Scale (EDSS), et al.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 18 years old;
2. Diagnosis of NMO or NMO spectrum disorder according to the 2015 International Panel for Neuromyelitis Optica Diagnosis criteria;
3. Clinical evidence of either at least one attack requiring rescue therapy (intravenous corticosteroids, intravenous immunoglobulin, plasma exchange, or a combination of these therapies) in the year before screening or at least two attacks requiring rescue therapy in the 2 years before screening;
4. EDSS <=6.0;
5. Patients were seropositive for AQP4-IgG;
6. Able and willing to give written informed consent and comply with the requirements of the study protocol.

Exclusion Criteria:

1. Current evidence or known history of clinically significant infection (Herpes simplex virus, varicella-zoster virus, cytomegalovirus, Epstein-Barr virus, human immunodeficiency virus, Hepatitis viruses, Syphilis, etc);
2. Participation in another interventional trial within the last 3 months Tumor disease currently or within last 5 years;
3. Pregnant, breastfeeding, or child-bearing potential during the course of the study Clinically relevant heart, liver, kidney or bone marrow function disorder.
4. Have a history of venous thromboembolism (VTE), or are considered at high risk for VTE by the investigator.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-04-15 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The number of attacks | From baseline to one year after
  An acute attack was defined as a new neurological worsening lasting for at least 24 hours and occurring more than 30 days after the previous attack

SECONDARY OUTCOMES:
Changes in EDSS | Changes in EDSS from baseline to 52 weeks
  The Expanded Disability Status Scale (EDSS) is a rating system that is frequently used for classifying and standardizing the severity and progression. EDSS ranges from 0 to 10.
Changes in the number of New, and/or Enlarging T2 Hyperintense Lesions as Detected by Optic nerve,brain and spinal cord Magnetic Resonance Imaging (MRI) | From baseline to 52 weeks
  The total number of new and/or enlarging T2 lesions for all participants was calculated as the sum of the individual number of lesions at Weeks 12, 24, and 52
Changes in peripheral blood B cell subsets | From baseline to 52 weeks
  Compare peripheral blood plasma cells before and one year after initial intervention
Changes in serum AQP4 antibodies | From baseline to 52 weeks
  Compare serum AQP4-ab titers before and one year after initial intervention
Incidence of treatment-emergent adverse events [safety and tolerability] | From baseline to 52 weeks
  Adverse events related to belimumab are recorded

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Liu, M.D.,PhD, Principal Investigator — Tianjin Medical University General Hospital
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality, China